CLINICAL TRIAL: NCT01894451
Title: Pilot Study of Zirconium-89 Bevacizumab Positron Emission Tomography for Imaging Angiogenesis in Patients With Inflammatory Breast Carcinoma Receiving Preoperative Chemotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather A. Jacene, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-147
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Inflammatory Breast Carcinoma
Keywords: Inflammatory Breast Carcinoma; 89Zr-bevacizumab
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — 89Zr-bevacizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-bevacizumab-PET/CT Scan (Experimental): * 89Zr-bevacizumab-PET/CT will be performed at baseline, after 2 cycles of preoperative chemotherapy, and at the completion of preoperative chemotherapy.
  * The 89Zr-bevacizumab-PET/CT imaging procedure is detailed in Appendix A and is briefly described below.
  Participants will be injected with 1 mCi of 89Zr-bevacizumab intravenously and PET/CT images will be obtained at 3-4 days after 89Zr-bevacizumab administration to allow time for antibody accumulation in the tumor. Imaging will be performed on a Centers for Quantitative Imaging Excellence (CQIE) qualified PET/CT scanner at the Dana-Farber Cancer Institute. After the baseline scan, subsequent scans will be obtained on the same PET/CT scanner for an individual participant.
  Interventions: Drug: 89Zr-bevacizumab; Procedure: FDG-PET/CT; Procedure: MRI scan; Procedure: Tumor biopsies

INTERVENTIONS:
Drug: 89Zr-bevacizumab — 89Zr-bevacizumab is a newly developed radiotracer. Radiotracers are compounds or drugs that are attached to small amounts of a radioactive substance. The amount of the compound or drug in a radiotracer is also very small. Radiotracers are used to make images of processes that are happening in the body, but they do not affect how the body works. 89Zr-bevacizumab is made up of the drug bevacizumab and the radioactive substance zirconium-89 (89Zr). 89Zr-bevacizumab is used for an imaging procedure called positron emission tomography/computed tomography (PET/CT). 89Zr-bevacizumab-PET/CT will be performed in this study at baseline, after 2 cycles of preoperative chemotherapy and at the completion of chemotherapy.
Procedure: FDG-PET/CT — FDG-PET/CT scan: Pictures of your organs will be taken using a PET (Positron Emission Tomography) scanner. At the same time, a CT (computed tomography) scan will be performed. FDG, a radioactive substance similar to glucose (or sugar), will be injected into your vein using a needle prior to performing the PET/CT scan. After the injection, you will be asked to sit quietly for one hour to let the FDG absorb into the body. After this hour, you will be asked to lie flat on your back for up to 50 minutes while the PET and CT images are being taken. This FDG-PET/CT scan is part of regular cancer care. If you have had this test within 14 days of study enrollment, you may or may not have to have this test repeated.
Procedure: MRI scan — • MRI Scan: MRI (Magnetic Resonance Imaging) scans of the breast will be taken. You will receive an injection of a dye before the MRI. You will be asked to lie flat on your back in the scanner for up to 30 minutes for pictures to be taken. This MRI scan is part of regular cancer care. If you have had this test within 14 days of study enrollment , you may or may not have to have this test repeated.
Procedure: Tumor biopsies — Tumor biopsies: Prior to starting your treatment, a radiologist will use breast MRI or ultrasound imaging to localize an area of your tumor in the breast for a research biopsy. The biopsy procedure is done in an outpatient setting using a done using a needle to obtain tissue. A local anesthetic will be given to minimize any pain; however, after the procedure you can expect some discomfort and possible bruising. This biopsy is part of research.

SUMMARY:
This research study is a pilot study, which tests the ability of an investigational compound to be used in humans for further studies. "Investigational" means that 89Zr-bevacizumab for PET/CT imaging is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved 89Zr-bevacizumab for PET/CT imaging for use in patients, including people with your type of cancer.

89Zr-bevacizumab is a newly developed radiotracer. Radiotracers are compounds or drugs that are attached to small amounts of a radioactive substance. The amount of the compound or drug in a radiotracer is also very small. Radiotracers are used to make images of processes that are happening in the body, but they do not affect how the body works. 89Zr-bevacizumab is made up of the drug bevacizumab and the radioactive substance zirconium-89 (89Zr). 89Zr-bevacizumab is used for an imaging procedure called positron emission tomography/computed tomography (PET/CT). This radiotracer has been used in other research studies. Information from those other research studies suggests that 89Zr-bevacizumab-PET/CT imaging may be able to measure new blood vessel formation to determine where the cancer is in your body and if your cancer is being killed by chemotherapy.

DETAILED DESCRIPTION:
Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about your health, current medications, and any allergies. This is part of regular cancer care.
* Physical exam, your doctor will examine your body, including measuring your height, weight, and vital signs (blood pressure, body temperature, pulse rate and breathing rate). This is part of regular cancer care.
* Blood tests (approximately 3 teaspoons) will be drawn for tests to check how well your organs are functioning. This is part of regular cancer care.
* Blood pregnancy test will be performed for women who can become pregnant. About 1 teaspoon of blood will be drawn for the blood pregnancy test. This is part of regular cancer care.
* Performance status, to see how you carry out your daily activities. This is done by talking with you. This is done as part of regular cancer care.

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

After the screening procedures confirm that you are eligible to participate in the research study:

Your primary oncologist will decide what chemotherapy you receive.

Before beginning preoperative chemotherapy (baseline):

Before beginning chemotherapy, you will undergo tests or procedures for the research study. Some of these tests and procedures are part of regular cancer care and some are being performed as part of the research study only.

* FDG-PET/CT scan: Pictures of your organs will be taken using a PET (Positron Emission Tomography) scanner. At the same time, a CT (computed tomography) scan will be performed. FDG, a radioactive substance similar to glucose (or sugar), will be injected into your vein using a needle prior to performing the PET/CT scan. After the injection, you will be asked to sit quietly for one hour to let the FDG absorb into the body. After this hour, you will be asked to lie flat on your back for up to 50 minutes while the PET and CT images are being taken. This FDG-PET/CT scan is part of regular cancer care. If you have had this test within 14 days of study enrollment, you may or may not have to have this test repeated.
* MRI Scan: MRI (Magnetic Resonance Imaging) scans of the breast will be taken. You will receive an injection of a dye before the MRI. You will be asked to lie flat on your back in the scanner for up to 30 minutes for pictures to be taken. This MRI scan is part of regular cancer care. If you have had this test within 14 days of study enrollment , you may or may not have to have this test repeated.
* 89Zr-bevacizumab-PET/CT Scan: More pictures of your organs will be taken using a PET (Positron Emission Tomography) scanner. At the same time, a CT (computed tomography) scan will be performed. 89Zr-bevacizumab will be injected into your vein using a needle. You will be observed for approximately 1 hour after the injection of 89Zr-bevacizumab. It takes 3 to 4 days for the 89Zr-bevacizumab to be absorbed into the body. Therefore, the research PET and research CT scans (89Zr-bevacizumab-PET/CT) will be performed 3 to 4 days after the 89Zr-bevacizumab is injected into your vein.
* This 89Zr-bevacizumab-PET/CT scan is part of research (in addition to the FDG-PET/CT scan) and is not part of regular cancer care.
* Vital signs, including heart rate, blood pressure, temperature, and respiratory rate, will be performed immediately before and then approximately 5, 30, and 60 minutes after injection of 89Zr-bevacizumab and just before 89Zr-bevacizumab-PET/CT imaging. This is part of research.
* Blood pregnancy test will be performed for women who can become pregnant. About 1 teaspoon of blood will be drawn for the blood pregnancy test. If your blood pregnancy test to determine if you could be in the study was done longer than 24 hours before the injection of 89Zr-bevacizumab, it will be repeated.
* Blood tests (approximately 3 teaspoons) will be drawn for tests to check how well your organs are functioning. This is part of regular cancer care.
* Tumor biopsies: Prior to starting your treatment, a radiologist will use breast MRI or ultrasound imaging to localize an area of your tumor in the breast for a research biopsy. The biopsy procedure is done in an outpatient setting using a done using a needle to obtain tissue. A local anesthetic will be given to minimize any pain; however, after the procedure you can expect some discomfort and possible bruising. This biopsy is part of research.

After 2 cycles of preoperative chemotherapy: Two to five days prior to starting your third cycle of chemotherapy, study tests and procedures will be performed. Some of these tests and procedures are part of regular cancer care and some are being performed as part of the research study only.

* FDG-PET/CT scan: The procedure is the same as that is described above. This FDG-PET/CT scan is part of research.
* MRI Scan: The procedure is the same as that is described above. This MRI scan is part of research.
* 89Zr-bevacizumab-PET/CT Scan: The procedure is the same as that is described above. This 89Zr-bevacizumab-PET/CT scan is part of research.
* Vital signs, including heart rate, blood pressure, temperature, and respiratory rate, is the same as that is described above. This is part of research.
* Blood pregnancy test will be performed for women who can become pregnant. This test is the same as that is described above. This is part of research.
* Blood tests (approximately 3 teaspoons) will be drawn for tests to check how well your organs are functioning. This is part of regular cancer care.
* Tumor biopsies: The procedure is the same that is described above. This biopsy is part of research.

After the completion of preoperative chemotherapy: Within 1-2 weeks after completing preoperative chemotherapy, study tests and procedures will be repeated to determine how well your cancer responded to the treatment. Some of these tests and procedures are part of regular cancer care and some are being performed as part of the research study only.

* FDG-PET/CT scan: The procedure is the same as that is described above. This FDG-PET/CT scan is part of research.
* MRI Scan: The procedure is the same as that is described above. This MRI scan is part of regular cancer care.
* 89Zr-bevacizumab-PET/CT Scan: The procedure is the same as that is described above. This 89Zr-bevacizumab-PET/CT scan is part of research.
* Vital signs, including heart rate, blood pressure, temperature, and respiratory rate, is the same as that is described above. This is part of research.
* Blood pregnancy test will be performed for women who can become pregnant. This test is the same as that is described above. This is part of research.
* Blood tests (approximately 3 teaspoons) will be drawn for tests to check how well your organs are functioning. This is part of regular cancer care.

Surgery: After completing preoperative chemotherapy, your primary oncologist and surgeon will determine if you are eligible to undergo breast surgery. Breast surgery is part of regular cancer care. During your surgery, tissue from your tumor will be removed and tested for how well your cancer responded to treatment. This is part of regular cancer care. If there is enough tissue available after the tissue has been tested for how well your tumor responded to treatment, some tissue will be taken for research. If you are not able to undergo breast surgery, then you will have a tumor biopsy similar to before starting and after 2 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Participants must have histologically or cytologically confirmed HER2 negative invasive breast adenocarcinoma.
* Participants must have clinical characteristics consistent with IBC, characterized by a rapid onset of clinical findings exemplified as diffuse edema and erythema of the breast, often without a palpable mass.
* Age ≥ 21 years. Because no dosing or adverse event data are currently available on the use of 89Zr-bevacizumab in participants <21 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* Any stage is eligible.
* Participants must be eligible for preoperative chemotherapy for IBC as determined by the treating physician.
* The effects of 89Zr-bevacizumab on the developing human fetus are unknown. For this reason and because radiopharmaceuticals may be teratogenic, women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability and willingness to comply with the study procedures.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must be willing to have research biopsies at baseline and after 2 cycles of preoperative chemotherapy, and possibly at the completion of preoperative chemotherapy.
* ECOG performance status ≤ 2.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:
* Pregnant women are excluded from this study because 89Zr-bevacizumab and 18F-FDG are radiopharmaceuticals with the potential for teratogenic effects. Because of the radiation exposure to a nursing infant from 89Zr-bevacizumab and 18F-FDG, women who are breastfeeding are also excluded from this study. In addition, bevacizumab may cause fetal harm based on animal studies (2).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery or significant bleeding episodes within 28 days before study initiation. Major surgery does not include: breast or other biopsies obtained for diagnosis, placement of radio-opaque clip to localize a tumor or tumors for subsequent surgical resection, placement of central venous access, pretreatment lymph node sampling. Significant bleeding episodes are defined for the purpose of this study as hemoptysis or upper/lower gastrointestinal bleeding.

Although bevacizumab will be administered in tracer quantities in this study and is not expected to have pharmacologic effects, participants with major surgery or significant bleeding episodes within 28 days before study initiation may be at a higher risk of bleeding.

Contraindications for MRI with contrast or PET/CT including:

* Cardiac pacemaker, implanted cardiac defibrillator, pacing wires, internal electrodes
* Aneurysm clips
* Cochlear, otologic, or other ear implant
* Tissue expander
* Swan-Ganz or Thermo Dilution
* Moderate renal insufficiency (estimated GFR less than 60 mL/min/1.73 m2) to end stage renal disease (estimated GFR less than 15 mL/min/1.73 m2 or a serum creatinine more than 3 mg/dL), who are not on dialysis, and patients with renal failure on chronic dialysis
* Severe claustrophobia
* History of multiple or severe allergic reactions attributed to immunoglobulins or MRI contrast agents.
* Any past or current condition that in the opinion of the study investigators would confound the results of the study or pose additional risk to the patient by their participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Quality Control Standards for Radiopharmamceuticals and Number of Successfully Acquired 89Zr-bevacizumab-PET/CT scans | 2 years
  In order to determine if 89Zr-bevacizumab-PET/CT scanning is feasible, we will determine results of radiolabeling of chelated bevacizumab including the radiolabeling yield, specific activity, and radiochemical purity and the number of successfully acquired 89Zr-bevacizumab-PET/CT scans.

SECONDARY OUTCOMES:
Number of related adverse events after the intravenous administration of 89Zr-bevacizumab. | 2 years
  To determine the safety of 89Zr-bevacizumab-PET/CT imaging in patients with IBC, the number of adverse events related to the radiotracer (89Zr-bevacizumab) will be determined.
Biodistribution of 89Zr-bevacizumab and individual organ and effective dose of 89Zr-bevacizumab | 2 Years
Amount of 89Zr-bevacizumab uptake in IBC tumor and measures of tumor angiogenesis in research biopsy specimens. | 2 Years
  The amount of 89Zr-bevacizumab uptake in IBC tumor will be primarily given by standardized uptake values from PET/CT imaging. Measures of tumor angiogenesis are intratumoral microvessel density (MVD), vessel diameter, and vascular pericyte coverage
Changes in tumor uptake of 89Zr-bevacizumab and FDG during and after preoperative chemotherapy and response in primary IBC tumor MRI. | 2 Years
  This outcome aims to determine if 89Zr-bevacizumab provides similar results in regards to monitoring therapy response compared to standard modalities, FDG-PET/CT and MRI breast
To correlate the changes in tumor uptake on 89Zr-bevacizumab-PET/CT with standard imaging response using MRI and FDG-PET/CT | 2 Years

OTHER OUTCOMES:
Visualization of primary IBC tumor and visualization and number of distant metastases | 2 years
  This is an exploratory outcome measure to see if 89Zr-bevacizumab detects primary and metastatic IBC tumor in a similar fashion
Percent change in 89Zr-bevacizumab tumor uptake in primary IBC tumor between the baseline and post preoperative chemotherapy PET/CT scans and residual cancer burden at mastectomy/tissue sampling if residual disease | 2 years
  This outcome measure is exploratory to investigate whether changes in tumor uptake of 89Zr-bevacizumab can predict response in mastectomy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Jacene, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts